CLINICAL TRIAL: NCT04277806
Title: Study on the New Feeding Protocol of Promoting Very Preterm Infants to Attain Full Oral Feeding Earlier
Brief Title: Promoting Full Oral Feeding in Preterm Infants Less Than 30 Weeks Gestational Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-298
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Preterm Infants

STUDY DESIGN:
Intervention Model Description: Randomized controlled study. Standard group: old protocol. Intervention group: New protocol.
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomized allocation was concealed in double-enclosed, opaque, sealed and sequentially numbered envelops and opened when the infant was found to be eligible by the neonatal team in the NICU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): No interventions would be conducted in this group and the preterm infants would be fed in the normal way.
- Intervention group (Experimental): The preterm infants in this group would be fed according to the new process.
  Interventions: Behavioral: New Oral feeding process

INTERVENTIONS:
Behavioral: New Oral feeding process — From the beginning of 32 weeks, try oral feeding once a day, suck pacifier for 10 minutes before feeding. When she/he can finish 50% of the amount of one meal in consecutive two days, and there is no adverse events happened, then we will try oral feeding twice a day. In the same way, in the oral feeding she/he can finish 50% of this meal in consecutive two days, there is no adverse events happened, then we will try three oral feedings three times a day. We wil continue the process until the infant can be fully oral fed by herself/himself.
  Arms: Intervention group

SUMMARY:
The investigators plan to use a new process to shorten the time of attaining full oral feeding in preterm infants less than 30 weeks gestational age.

DETAILED DESCRIPTION:
In the neonatal intensive care unit, the attention of oral feeding of premature infants is far less than that of mechanical ventilation, antibiotics and other medical treatment, the use of parenteral nutrition, etc., and it is often not until the premature infants are enough mature and stable, or even before discharge that the caregivers pay attention to the problem of oral feeding. At this time, the corrected gestational age of premature infants is almost 36 weeks, but in fact the study shows that preterm infants have the ability of self feeding when they are about 32 weeks old. And oral feeding is very helpful to improve their nutritional status, reduce the use of parenteral nutrition and other forms of enteral nutrition, prevent complications and shorten the length of stay. Therefore, this study plans to use a new process to promote oral feeding and to verify whether it is feasible to earlier attainment of full oral feeding in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age less than 30 weeks
* The parents are positive to treat the infants

Exclusion Criteria:

* Fetal edema
* Very critical with OI more than 40
* Apgar score less than 5 at ten minutes after birth
* The parents refuse to treat the infants
* Severe IVH (more than grade IV )
* PVL
* Died before oral feeding starts

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Age at full oral feeding | During the procedure
  Days of life when the infant attain full oral feeding among two groups.

SECONDARY OUTCOMES:
The length of hospital stay | During the procedure
  The length of hospital stay of participates in two groups.
Incidence of complications | During the procedure
  Complications include NecrotizingEnterocolitis，any infections，Intraventricular hemorrhage，Bronchopulmonary dysplasia，etc. The variables of complications will be set to 1 as any symptoms mentioned above appeared during the hospitalization and none for 0. The incidence would be calculated in two groups.
Corrected gestational age at full oral feeding | During the procedure
  Corrected gestational age when the infant attain full oral feeding among two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China